CLINICAL TRIAL: NCT04639609
Title: Characterization of Neuromuscular Function and Fatigue After Breast Cancer Treated With Adjuvant Chemotherapy
Brief Title: Characterization of Neuromuscular Function and Fatigue After Breast Cancer Treated With Adjuvant Chemotherapy (PROTECT-04)
Acronym: PROTECT-04
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Collaborators: UR 3072 - Mitochondrie, Stress oxydant et Protection musculaire (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-007; 2020-A01272-37 (Other: IDRCB)
Record Dates: First submitted 2020-11-02; First posted 2020-11-20 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 : Patients (Experimental)
  Interventions: Other: Characterization of Neuromuscular Function and Fatigue
- Group 2 : healthy volunteers (Other)
  Interventions: Other: Characterization of Neuromuscular Function and Fatigue

INTERVENTIONS:
Other: Characterization of Neuromuscular Function and Fatigue — at inclusion

SUMMARY:
This is a transversal monocentric study comparing two groups of women (group 1, patient group : patients who have been treated for a breast cancer with taxane-based chemotherapy ; group 2, control group : healthy volunteers). The aim of this study is to evaluate if a difference exists regarding the maximal isometric muscle strength between group 1 and 2.

DETAILED DESCRIPTION:
All subjects will be evaluated a single time during two hours. For patients from group 1 the evaluation should take place within the two weeks that follow the end of adjuvant treatment. There is no specificity regarding evaluation of volunteers from group 2, their evaluation can take place at any time.

ELIGIBILITY:
Inclusion Criteria :

Group 1 - Patients :

* Give written inform consent
* Age ≥ 18 years
* Affiliate to social security system
* Ability to speak, understand and read French
* Breast cancer, Stage II or III, treated by taxane-based chemotherapy

Group 2 - Control group :

* Give written inform consent
* Age ≥ 18 years
* Affiliate to social security system
* Ability to speak, understand and read French

Exclusion Criteria:

Group 1 - Patients :

* < 18 years old or patients ≥ 18 years old under guardianship, or supervision
* Psychiatric, musculoskeletal or neurologic disorders
* Patients presenting one of the following contraindications to transcranial magnetic stimulation :
* Presence of a implanted metallic foreign-body (cochlear implant, drug pump system, pacemaker, etc.)
* History of epilepsy
* Brain injury (vascular, traumatic, tumour-induced, infectious or metabolic)
* Women that are pregnant
* Serious or recent heart disease

Group 2 -Control group :

* < 18 years old or patients ≥ 18 years old under guardianship, or supervision
* Psychiatric, musculoskeletal or neurologic disorders
* Pacemaker implantation
* History of cancer
* All known chronic disease
* Subjects presenting one of the following contraindications to transcranial magnetic stimulation :
* Presence of a implanted metallic foreign-body (cochlear implant, drug pump system, pacemaker, etc.)
* History of epilepsy
* Brain injury (vascular, traumatic, tumour-induced, infectious or metabolic)
* Women that are pregnant
* Serious or recent heart disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
Maximal isometric muscle strength for knee extensors | At Inclusion
  Measured with force sensors. Significant differences between the two groups will be assessed

SECONDARY OUTCOMES:
Number of Participants with neuromuscular fatigue | At Inclusion
  Assessment using surface electromyography. Significant differences between the two groups will be assessed.
Number of Participants with neuromuscular fatigue | At Inclusion
  Assessment using percutaneous electric nerve stimulation. Significant differences between the two groups will be assessed.
Number of Participants with neuromuscular fatigue | At Inclusion
  Assessment using transcranial magnetic stimulation. Significant differences between the two groups will be assessed.
Number of Participants with subjective fatigue. | At Inclusion
  Questionnaire Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-F) version 4.
  Significant differences between the two groups will be assessed.
Number of Participants with muscle architecture. | At Inclusion
  Assessment using muscle ultrasonography. Significant differences between the two groups will be assessed.
Number of Participants with body composition. | At Inclusion
  Assessment using bio-impedance analysis. Significant differences between the two groups will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Cancerologie Strasbourg Europe, Strasbourg, France

REFERENCES:
- [Derived] Hucteau E, Mallard J, Pivot X, Schott R, Pflumio C, Trensz P, Favret F, Pagano AF, Hureau TJ. Exacerbated central fatigue and reduced exercise capacity in early-stage breast cancer patients treated with chemotherapy. Eur J Appl Physiol. 2023 Jul;123(7):1567-1581. doi: 10.1007/s00421-023-05177-5. Epub 2023 Mar 20. PMID 36939876